CLINICAL TRIAL: NCT04372771
Title: Comparison of Two Diet and Exercise Approaches on Weight Loss and Health Outcomes in Obese Women
Brief Title: Comparing Diet and Exercise Approaches in Women
Acronym: CWW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Responsible Party: Principal Investigator, Richard B. Kreider, Executive Director, Human Clinical Research Facility, Texas A&M University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IRB2010-0130F
Record Dates: First submitted 2020-04-30; First posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Diet Modification
Keywords: Exercise Intervention

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No diet or exercise intervention
- Curves Program (Experimental): The Curves group will follow the high protein/low fat diet (30% carbohydrate, 45% protein, 25% fat) for 7-days at 1,200 kcals/day and then 1,500 kcals/day for the remaining 21-days of the 30-day diet period. The participants will then consume a normal maintenance diet (2,200 kcals/d; 45% carbohydrate, 30% protein, 25% fat) for 30-days. During the maintenance period, participants will diet for 2-days at 1,200 kcals/day if they gain 3 pounds of weight.
  Interventions: Other: Curves Circuit
- Weight Watchers Momentum Program (Experimental): This program is based on the Weight Watchers four pillar approach (food, exercise, behavior and support). The Momentum Program uses POINTS values to help keep track of what you eat. A POINTS "budget" will be personalized for you at the weekly meetings.
  Interventions: Other: Weight Watchers

INTERVENTIONS:
Other: Curves Circuit — The Curves Circuit consists performing 13 hydraulic resistance exercise machines that utilize bidirectional resistance that work all major muscle groups. These are interspersed with floor-based calisthenic exercises designed to maintain an elevated heart rate.
  Arms: Curves Program
Other: Weight Watchers — The Weight Watchers program encourages one to increase physical activity.
  Arms: Weight Watchers Momentum Program

SUMMARY:
The purpose of this study is to determine whether following a Curves high protein/low fat diet (30% carbohydrate, 45% protein, 25% fat) for 30-days several times during 16 weeks of participating in the Curves fitness program promotes stepwise reductions in body weight, improvements in body composition and/or improvements in markers of fitness and health better than following the Weight Watchers Momentum Program for the same time period.

DETAILED DESCRIPTION:
The Curves International fitness and weight loss program has become a very popular means of promoting health and fitness among women. The program involves a 30-minute circuit training program and a weight management program involving periods of moderate caloric restriction (1,200 to 1,600 calories per day) followed by short periods of higher caloric intake (2,600 calories per day). The program is designed to promote a gradual reduction in body fat while increasing strength and muscle mass/tone. Researchers in the Exercise and Sport Nutrition Lab at Texas A&M University have conducted an extensive study on the effectiveness and safety of the Curves fitness and diet program. Results of this initial study have shown that the program promotes weight loss, improves markers of health, and improves fitness. The Weight Watchers program is another popular weight loss program. It provides a systematic approach to diet and exercise throughout the weight-loss process. Consequently we are interested in comparing the efficacy of both programs to one another. The purpose of this study is to determine whether following a Curves high protein/low fat diet (30% carbohydrate, 45% protein, 25% fat) for 30-days several times during 16 weeks of participating in the Curves fitness program promotes stepwise reductions in body weight, improvements in body composition and/or improvements in markers of fitness and health better than following the Weight Watchers Momentum Program for the same time period.

ELIGIBILITY:
Inclusion Criteria:

* Participant is female
* Participant is between the ages of 18 and 45
* Participant is sedentary and overweight (BMI > 27)

Exclusion Criteria:

* Participant has any metabolic disorder including known electrolyte abnormalities, heart disease, arrhythmias, diabetes, thyroid disease, or hypogonadism;
* Participant has a history of hypertension, hepatorenal, musculoskeletal, autoimmune or neurological disease;
* Participant is taking thyroid, hyperlipidemic, hypoglycemic, anti-hypertensive or androgenic medications;
* Participant has been pregnant or lactating within the past 12 months or are planning to become pregnant during the next 12 months;
* Participant is involved in a planned exercise program (> 30 min./d. 3 d./wk.) within 3 - 6 months prior to the start of the study;
* Participant has taken any weight loss medications and/or dietary supplements that may affect muscle mass or body weight during the three month time period prior to beginning the study;
* Participant has a recent history of weight change (+/- 7 lbs. within the last 3 months).

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-04-19 (Actual); Primary Completion 2012-03-22 (Actual); Study Completion 2012-03-22 (Actual)

PRIMARY OUTCOMES:
Body Composition: Body Weight | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in body weight (lbs. body weight) obtained via digital scale and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Fat Mass | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in body composition (lbs. fat mass) obtained via Dual-Energy X-Ray Absorptiometry (DXA) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Lean Mass | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in body composition (lbs. lean mass) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Body Composition: Percent Body Fat | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in body composition (% body fat) obtained via DXA and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Energy Homeostasis: Resting Energy Expenditure (REE) | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in REE obtained via metabolic cart and expressed in absolute (kcal/d) and relative terms (kcals/kg/d) and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)

SECONDARY OUTCOMES:
Muscular Strength: 1 Repetition Maximum (1 RM) Bench Press | Measured prior to supplementation (Pre), and after 16 weeks
  Changes in bench press 1 Repetition Maximum (1RM) obtained from a bench press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Strength: 1 Repetition Maximum (1 RM) Leg Press | Measured prior to supplementation (Pre), and after 16 weeks
  Changes in leg press 1RM obtained from a leg press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Endurance: 80% of 1 Repetition Maximum (1 RM) Bench Press Endurance Test | Measured prior to supplementation (Pre), and after 16 weeks
  Changes in total repetitions at 80% of 1RM obtained from a bench press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Muscular Endurance: 80% of 1 Repetition Maximum (1 RM) Leg Press Endurance Test | Measured prior to supplementation (Pre), and after 16 weeks
  Changes in total repetitions at 80% of 1RM obtained from a leg press test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: Cholesterol | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: HDL Cholesterol | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in HDL cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: LDL Cholesterol | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in LDL cholesterol obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: Triglycerides | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in triglycerides obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Lipid Panel: Cholesterol:HDL Ratio | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in cholesterol to HDL cholesterol ratio obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Comprehensive Metabolic Panel (CMP): Glucose | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in glucose obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hormones: Insulin | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in insulin obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hormones: Leptin | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in leptin obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR): Homeostatic Model Assessment of Insulin Resistance | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in HOMA-IR obtained via venous blood draws and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Heart Rate (HR) | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in resting heart rate (HR) obtained via a blood pressure meter and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Systolic Blood Pressure (SBP) | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in resting systolic blood pressure (SBP) obtained via a blood pressure meter and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Hemodynamic Variable: Resting Diastolic Blood Pressure (SBP) | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in resting diastolic blood pressure (DBP) obtained via a blood pressure meter and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Waist Circumference | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in waist circumference obtained via tape measure and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Hip Circumference | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in hip circumference obtained via tape measure and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Anthropometric Measures: Waist to Hip Ratio | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in the ratio of waist to hip (waist/hip circumference) analyzed with related anthropometric outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Exercise Capacity: Peak Exercise Capacity (VO2) | Measured prior to supplementation (Pre), and after 16 weeks
  Changes in exercise capacity (VO2 max) obtained via a treadmill test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Exercise Capacity: Time to Peak Exercise Capacity (time to peak VO2) | Measured prior to supplementation (Pre), and after 16 weeks
  Changes in exercise capacity (time to peak VO2 max) obtained via a treadmill test and analyzed by General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Dietary Energy Intake: Total Caloric Intake (kcals/d) | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in caloric/energy intake (kcals/d) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Dietary Energy Intake: Carbohydrate | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in dietary carbohydrate intake (g/d and g/kg/d) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Dietary Energy Intake: Fat | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in dietary fat intake (g/d and g/kg/d) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)
Dietary Energy Intake: Protein | Measured prior to supplementation (Pre), and after 4, 6, 10, 12 and 16 weeks
  Changes in dietary protein intake (g/d and g/kg/d) analyzed with related energy intake outcome measures via General Linear Model multivariate and univariate analyses with repeated measures and mean change from baseline with 95% confidence intervals (CI's)

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Kreider, PhD, Principal Investigator — Texas A&M University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lockard B, Mardock M, Oliver JM, Byrd M, Simbo S, Jagim AR, Kresta J, Baetge CC, Jung YP, Koozehchian MS, Khanna D, Rasmussen C, Kreider RB. Comparison of Two Diet and Exercise Approaches on Weight Loss and Health Outcomes in Obese Women. Int J Environ Res Public Health. 2022 Apr 17;19(8):4877. doi: 10.3390/ijerph19084877. PMID 35457744